CLINICAL TRIAL: NCT01462227
Title: The Effect of Opiate Blockade With Naltrexone on Counterregulatory Mechanisms in Hypoglycemia
Brief Title: Effect of Naltrexone on Counterregulatory Mechanisms in Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HIC1006006927
Record Dates: First submitted 2011-10-26; First posted 2011-10-31 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia; Type 1 diabetes
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone (higher dose) (Experimental): Naltrexone 100mg tablets were randomly given on 1 of 2 occassions (the other was placebo). The drug was administered 12 hours and 1 hour orally pre-procedure to participants. Placebo was given to the high dose group on 1 of their 2 visits- the order in which placebo was given was randomized by dosage arm.
  Interventions: Drug: Naltrexone High Dose
- Naltrexone (lower dose) (Experimental): Naltrexone 50mg tablets were randomly given on 1 of 2 occassions (the other was placebo). The drug was administered 12 hours and 1 hour orally pre-procedure to participants. Placebo was given to the low dose group on 1 of their 2 visits- the order in which placebo was given was randomized by dosage arm.
  Interventions: Drug: Naltrexone Low Dose

INTERVENTIONS:
Drug: Naltrexone High Dose — Naltrexone 100mg for two administrations.
  Arms: Naltrexone (higher dose)
Drug: Naltrexone Low Dose — Naltrexone 50mg for two administrations.
  Arms: Naltrexone (lower dose)

SUMMARY:
Insulin treatment often causes the blood glucose levels to fall too low. The body usually responds to low blood glucose levels by releasing hormones which act against the insulin to help correct the low blood glucose levels. However, this hormone response can be altered in people with diabetes. Currently there are no therapeutic agents that can be used to improve the recovery from hypoglycemia (low blood sugar). Naltrexone is a tablet used to help people who are addicted to alcohol or morphine-based drugs to remain drug and alcohol-free but it can also affect the levels of the hormones which are released during hypoglycemia. The aim of this study is to determine whether naltrexone can be used to improve and accelerate the recovery from hypoglycemia in patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes (well controlled, 2-3 hypoglycemic episodes/wk) age 18-55, BMI 18-35

Exclusion Criteria:

* pregnancy
* significant diabetes complications
* liver disease, cirrhosis
* cardiac disease
* neurological disorder
* autonomic neuropathy
* kidney disease
* lactose intolerance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone (Lower Dose) First /Placebo Second: Naltrexone 50 mg, 1 tablet given 12 hours prior to visit orally Placebo given at time of visit orally
- Placebo First/ Naltrexone (Lower Dose) Second: Placebo given given 12 hours prior to visit orally Naltrexone 50 mg (1 tablet) given at time of visit orally
- Naltrexone (Higher Dose) First /Placebo Second: Naltrexone 100 mg, 1 tablet given 12 hours prior to visit orally Placebo given at time of visit orally
- Placebo First / Naltrexone (Higher Dose) Second: Placebo given 12 hours prior to visit orally Naltrexone 100 mg (1 tablet) given at time of visit orally
Period: First Assignment
Arm/Group | Naltrexone (Lower Dose) First /Placebo Second | Placebo First/ Naltrexone (Lower Dose) Second | Naltrexone (Higher Dose) First /Placebo Second | Placebo First / Naltrexone (Higher Dose) Second
Started | 4 | 2 | 6 | 5
Completed | 4 | 2 | 6 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Second Assignment
Arm/Group | Naltrexone (Lower Dose) First /Placebo Second | Placebo First/ Naltrexone (Lower Dose) Second | Naltrexone (Higher Dose) First /Placebo Second | Placebo First / Naltrexone (Higher Dose) Second
Started | 4 | 2 | 6 | 5
Completed | 3 | 1 | 5 | 5
Not Completed | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population includes subjects that completed study
Groups:
- Naltrexone (Lower Dose): Naltrexone: Naltrexone 50 mg, 1 tablet given every 12 hours orally
- Naltrexone (Higher Dose): Naltrexone: Naltrexone 100mg, 1 tablet given every 12 hours orally
- Total: Total of all reporting groups
Arm/Group | Naltrexone (Lower Dose) | Naltrexone (Higher Dose) | Total
Number analyzed (Participants) | 4 | 10 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (11) | 32.4 (12) | 32.4 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Glucose (mg/dL)
Description: Glucose was measured in the blood throughout the hyperinsulinemic-hypoglycemic clamp study.
Time Frame: End of study (up to 240 minutes)
Population: Subjects' data were pooled and only those that completed both visits are analyzed here.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Naltrexone (Lower Dose): Subjects were randomized to receive either Naltrexone 50 mg or placebo: 1 tablet given 12 hours prior to visit orally and again at time of visit.
- Naltrexone (Higher Dose): Subjects were randomized to receive either Naltrexone 100 mg or placebo: 1 tablet given 12 hours prior to visit orally and again at time of visit.
Arm/Group | Naltrexone (Lower Dose) | Naltrexone (Higher Dose)
Number analyzed (Participants) | 4 | 10
mg/dL
  Active Drug | 56.5 (3.7) | 52.8 (8.6)
  Placebo | 55.0 (2.8) | 52.8 (8.6)

2. Primary Outcome: Glucose Infusion Rate (mg/kg.Min)
Description: The glucose infusion rate corresponds to the amount of 20% dextrose given during the hyperinsulinemic-hypoglycemic clamp study, necessary to keep blood glucose levels at the target range (50-55 mg/dL).
Time Frame: End of study (up to 240 minutes)
Population: Subjects' data were pooled and only those that completed both visits are analyzed here.
Measure: Mean (Standard Deviation); unit: mg/kg.min
Arm/Group | Naltrexone (Lower Dose) | Naltrexone (Higher Dose)
Number analyzed (Participants) | 4 | 10
mg/kg.min
  Active Drug | 4.6 (2.7) | 6.3 (2.4)
  Placebo | 4.8 (4.0) | 5.9 (2.7)

3. Secondary Outcome: Glucagon (pg/mL)
Description: Glucagon was measured in the blood throughout the hyperinsulinemic-hypoglycemic clamp study.
Time Frame: End of study (up to 240 minutes)
Population: Subjects' data were pooled and only those that completed both visits are analyzed here.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Naltrexone (Lower Dose) | Naltrexone (Higher Dose)
Number analyzed (Participants) | 4 | 10
pg/mL
  Active Drug | 44.1 (17.4) | 48.9 (16.5)
  Placebo | 40.4 (7.9) | 53.6 (16.4)

4. Secondary Outcome: Cortisol (ug/dL)
Description: Cortisol was measured in the blood throughout the hyperinsulinemic-hypoglycemic clamp study.
Time Frame: End of study (up to 240 minutes)
Population: Subjects' data were pooled and only those that completed both visits are analyzed here.
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Naltrexone (Lower Dose) | Naltrexone (Higher Dose)
Number analyzed (Participants) | 4 | 10
ug/dL
  Active Drug | 22.9 (8.3) | 16.4 (8.1)
  Placebo | 16.0 (7.0) | 15.2 (5.2)

5. Secondary Outcome: Epinephrine (pg/mL)
Description: Epinephrine was measured in the blood throughout the hyperinsulinemic-hypoglycemic clamp study.
Time Frame: End of study (up to 240 minutes)
Population: Subjects' data were pooled and only those that completed both visits are analyzed here.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Naltrexone (Lower Dose) | Naltrexone (Higher Dose)
Number analyzed (Participants) | 4 | 10
pg/mL
  Active Drug | 92.75 (30.6) | 126.1 (98.0)
  Placebo | 42.75 (23.1) | 77.9 (65.8)

6. Secondary Outcome: Norepinephrine (pg/mL)
Description: Norepinephrine was measured in the blood throughout the hyperinsulinemic-hypoglycemic clamp study.
Time Frame: End of study (up to 240 minutes)
Population: Subjects' data were pooled and only those that completed both visits are analyzed here.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Naltrexone (Lower Dose) | Naltrexone (Higher Dose)
Number analyzed (Participants) | 4 | 10
pg/mL
  Active Drug | 248.3 (80.2) | 200.1 (77.4)
  Placebo | 282.8 (97.3) | 217.1 (91.5)

ADVERSE EVENTS:
Time Frame: End of study, up to 240 minutes.
Groups:
- Naltrexone (50 mg): Naltrexone 50 mg, 1 tablet given 12 hours and again at 1 hour prior to testing (orally).
- Placebo (Lower Dose Group); Placebo (Higher Dose): Placebo 1 tablet given 12 hours and again at 1 hour prior to testing (orally).
- Naltrexone (100 mg): Naltrexone 100 mg, 1 tablet given 12 hours and again at 1 hour prior to testing (orally).
Arm/Group | Naltrexone (50 mg) | Placebo (Lower Dose Group) | Naltrexone (100 mg) | Placebo (Higher Dose)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 5/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (50 mg) (N=4) | Placebo (Lower Dose Group) (N=4) | Naltrexone (100 mg) (N=10) | Placebo (Higher Dose) (N=10)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes